CLINICAL TRIAL: NCT04201405
Title: A Phase I-II, Study of Autologous CD34+ Haematopoietic Stem Cells Transduced Ex Vivo with CD11b Lentiviral Vector Encoding for Human SGSH in Patients with Mucopolysaccharidosis Type IIIA (MPS IIIa, Sanfilippo Syndrome Type A)
Brief Title: Gene Therapy with Modified Autologous Hematopoietic Stem Cells for Patients with Mucopolysaccharidosis Type IIIA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Orchard Therapeutics (Industry); CTI Clinical Trial and Consulting Services (Other); University College, London (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Rob Wynn, Professor, Manchester University NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R119861
Record Dates: First submitted 2019-12-05; First posted 2019-12-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Mucopolysaccharidosis Type IIIA
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haematopoietic stem cell gene therapy for MPS IIIA (Experimental): Open label
  Interventions: Drug: Autologous CD34+ cells transduced with a lentiviral vector containing the human SGSH gene

INTERVENTIONS:
Drug: Autologous CD34+ cells transduced with a lentiviral vector containing the human SGSH gene — Autologous CD34+ haematopoietic stem cells from MPS IIIA patients will be genetically modified ex vivo using CD11b.SGSH Lentiviral vector (LV), a self-inactivating LV expressing the SGSH gene codon optimized for human use and regulated by a human CD11b myeloid-specific promoter. Cells will be cryopreserved prior to patient administration.

SUMMARY:
Patients with MPS IIIA have a clinical disorder marked by severe and progressive brain disease and neurological symptoms due to the accumulation of undigested glycosaminoglycans in all cells of the body.

This study will be the first in human clinical trial to explore the safety, tolerability and clinical efficacy of ex vivo gene therapy (autologous CD34+ cells transduced with a lentiviral vector containing the human SGSH gene) in MPSIIIA patients. Following treatment with the gene therapy patients will be followed up for a minimum of 3 years.

DETAILED DESCRIPTION:
MPS IIIA is caused by a deficiency of the heparan-N-sulfatase (SGSH) enzyme, leading to the accumulation of the glycosaminoglycan heparan sulphate in the lysosomes. Untreated patients of MPS IIIA experience rapid and progressive neurologic deterioration. To date, there is no effective disease-modifying treatment for patients suffering from MPS IIIA.

This study aims to recruit 3 to 5 patients with MPS IIIA who satisfy the inclusion and exclusion criteria and provide full consent, between 3 months and 24 months of age. The investigational medicinal product (IMP) will be a cell-based gene therapy that uses genetically modified autologous CD34+ haematopoietic stem cells transduced with a lentiviral vector containing the human SGSH gene. Patients will be followed up for a minimum of 3 years after gene therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of a legally authorized guardian(s)
2. Age at baseline ≥3 months and ≤24 months
3. Normal cognitive function or mild cognitive deterioration (subject has a Development Quotient (DQ) score ≥80) at baseline as determined by the Bayley Scale of Infant Development-third edition (BSID-III), cognitive domain)
4. Sibling or relative of known MPS IIIA patients with rapidly progressing phenotype, or genotype associated with rapidly progressing phenotype, or presence of somatic features predictive of rapid progression
5. SGSH activity ≤10% of the Lower Limit of Normal as measured in leukocytes, plus either (1) a normal enzyme activity level of at least one other sulfatase (to rule out multiple sulfatase deficiency) as measured in leukocytes or (2) two documented mutations in the SGSH gene.
6. Medically stable and able to accommodate the protocol requirements, including travel without placing an undue burden on the patient/patient's family, as determined by the CI.

Exclusion Criteria:

1. The subject has received stem cell, gene therapy or enzyme replacement therapy (any route of administration)
2. Subject currently enrolled in other interventional clinical trials.
3. Contraindications for MRI scans.
4. The subject has a history of poorly controlled seizures.
5. Homozygous or compound heterozygous for the S298P mutation or any other mutation known to be associated to slow-progressing phenotype.
6. The subject is currently receiving psychotropic or other medications which, in the CI's opinion, would be likely to substantially confound test results.
7. The subject has received any investigational medicinal product (including Genistein) within 30 days prior to the Baseline visit or is scheduled to receive any investigational medicinal product during the course of the study.
8. Documented Human Immunodeficiency Virus (HIV) infection (positive HIV RNA and/or anti-p24 antibodies).
9. Malignant neoplasia (except local skin cancer) or a documented history of hereditary cancer syndrome. Subjects with a prior successfully treated malignancy and a sufficient follow-up to exclude recurrence (based on oncologist opinion) can be included after discussion and approval by the Medical Monitor.
10. Myelodysplasia, cytogenetic alterations characteristic of myelodysplastic syndrome and acute myeloid leukaemia, or other serious haematological disorders.
11. The subject has a medical condition or extenuating circumstance that, in the opinion of the CI, might compromise the subject's ability to comply with protocol requirements, the subject's well-being or safety, or the interpretability of the subject's clinical data.
12. Visual or hearing impairment sufficient to preclude cooperation with neurodevelopmental testing.
13. Severe behavioural disturbances due to reasons other than MPS IIIA and likely to interfere with protocol compliance, as determined by the CI.
14. Known sensitivity to busulfan.
15. The receipt of live vaccinations within 30 days prior to study start.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability of the IMP in MPS IIIA patients: scale | up to 3 years
  Adverse events will be recorded and graded according to an adapted Pediatric Clinical Toxicity Scale from the National Institute Allergy and Infectious Diseases (NIAID), Autoimmuno-deficiency Syndrome (AIDS) Division
To evaluate the biological efficacy of IMP post-treatment: expression of SGSH in total leukocytes | 12 months post gene therapy
  Measured by the expression of SGSH in total leukocytes within or above normal range at 12 months post-IMP treatment
To assess the safety of the IMP in MPS IIIA patients | up to 3 years
  Presence of replication competent virus and integration events in the leukocytes

SECONDARY OUTCOMES:
To evaluate overall survival | up to 3 years
  Overall survival at 36 months post IMP administration compared to natural history data
To evaluate peripheral engraftment of the IMP | within 42 days of treatments
  Measured as absence of engraftment failure or delayed hematological reconstitution within the first 6 weeks of IMP delivery. Defined as three independent and consecutive days with absolute Neutrophil Count (ANC) >500/mm3 and/or Platelets >20,000/mm3 without transfusions, and/or Hb >8.0 g/dL without transfusions.
Change in adaptive behaviour | up to 3 years (multiple visits)
  Measured using the Vineland Adaptive Behaviour scales against natural history of MPSIIIA
Change in cognitive function | up to 3 years (multiple visits)
  Measurement of cognitive score (standard scores, age equivalent scores and development quotient) using the Bayley Scales of Infant Development, 3rd Edition [BSID-III] or Kaufman Assessment Battery for Children, 2nd Edition [KABC-II] against natural history of MPSIIIA
Change in patient behaviour | up to 3 years
  Measured using the Sanfilippo Behaviour Rating Scale against natural history of MPSIIIA
Change in patient quality of life | Up to 3 years
  Measured using the Infant Toddler Quality of Life questionnaire against natural history of MPSIIIA
Change in patient's daily living | Up to 3 years
  Measured using the Children sleep Questionnaire against natural history data

OTHER OUTCOMES:
To evaluate the effect of the IMP on heparan sulphate concentration in cerebrospinal fluid (CSF), plasma and urine | 6 months and 12 months post-IMP treatments and multiple other visits over time
  Measure change in ng/ml glycosaminoglycans in CSF from baseline following IMP administration
To evaluate the effect of the IMP on SGSH activity in CSF, plasma and peripheral blood mononuclear cells. | 6 months and 12 months post-IMP treatments and multiple other visits over time
  Change in SGSH activity measured from baseline
To evaluate clinical efficacy of the IMP on brain imaging biomarkers | up to 3 years
  Measure change in brain volume (total brain, grey and white matter, ventricle volume) by MRI and compare to baseline and natural history data to help assess brain development
To explore the presence of anti-SGSH antibodies following treatment with the IMP | up to 3 years
  Measure whether an immune response is generated against the SGSH enzyme

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bigger, Principal Investigator — The University of Manchester; Robert Wynn, Principal Investigator — MFT
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No, there is not a plan to make IPD available.

REFERENCES:
- [Background] Ellison SM, Liao A, Wood S, Taylor J, Youshani AS, Rowlston S, Parker H, Armant M, Biffi A, Chan L, Farzaneh F, Wynn R, Jones SA, Heal P, Gaspar HB, Bigger BW. Pre-clinical Safety and Efficacy of Lentiviral Vector-Mediated Ex Vivo Stem Cell Gene Therapy for the Treatment of Mucopolysaccharidosis IIIA. Mol Ther Methods Clin Dev. 2019 Apr 6;13:399-413. doi: 10.1016/j.omtm.2019.04.001. eCollection 2019 Jun 14. PMID 31044143
- [Background] Holley RJ, Wood SR, Bigger BW. Delivering Hematopoietic Stem Cell Gene Therapy Treatments for Neurological Lysosomal Diseases. ACS Chem Neurosci. 2019 Jan 16;10(1):18-20. doi: 10.1021/acschemneuro.8b00408. Epub 2018 Aug 23. PMID 30136572
- [Background] Ghosh A, Shapiro E, Rust S, Delaney K, Parker S, Shaywitz AJ, Morte A, Bubb G, Cleary M, Bo T, Lavery C, Bigger BW, Jones SA. Recommendations on clinical trial design for treatment of Mucopolysaccharidosis Type III. Orphanet J Rare Dis. 2017 Jun 26;12(1):117. doi: 10.1186/s13023-017-0675-4. PMID 28651568
- [Background] Sergijenko A, Langford-Smith A, Liao AY, Pickford CE, McDermott J, Nowinski G, Langford-Smith KJ, Merry CL, Jones SA, Wraith JE, Wynn RF, Wilkinson FL, Bigger BW. Myeloid/Microglial driven autologous hematopoietic stem cell gene therapy corrects a neuronopathic lysosomal disease. Mol Ther. 2013 Oct;21(10):1938-49. doi: 10.1038/mt.2013.141. Epub 2013 Jun 7. PMID 23748415
- [Background] Langford-Smith A, Wilkinson FL, Langford-Smith KJ, Holley RJ, Sergijenko A, Howe SJ, Bennett WR, Jones SA, Wraith J, Merry CL, Wynn RF, Bigger BW. Hematopoietic stem cell and gene therapy corrects primary neuropathology and behavior in mucopolysaccharidosis IIIA mice. Mol Ther. 2012 Aug;20(8):1610-21. doi: 10.1038/mt.2012.82. Epub 2012 May 1. PMID 22547151